CLINICAL TRIAL: NCT04491799
Title: Fecal Calprotectin Level in Differentiating Between Inflammatory and Non-inflammatory Diarrhea in Patients With Nosocomial Diarrhea
Brief Title: Fecal Calprotectin Level in Patients With Nosocomial Diarrhea
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Assist.Professor, Mahidol University
Other Study IDs: Si056/2019
Record Dates: First submitted 2020-04-26; First posted 2020-07-29 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Diarrhea; Calprotectin
Keywords: Nosocomial diarrhea; Fecal calprotectin
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool examination Stool C.difficile toxin Fecal calprotectin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nosocomial diarrhea: Patients who are hospitalized and develop diarrhea after 72 hours of hospitalization.
  Interventions: Diagnostic Test: Fecal calprotectin

INTERVENTIONS:
Diagnostic Test: Fecal calprotectin — Fecal calprotectin is a protein found in human neutrophils, and it is released during active periods of inflammation of intestine. The sensitivity and specificity has been reported at 93% and 96%, respectively in differentiating inflammatory bowel disease from irritable bowel syndrome in outpatient setting.

SUMMARY:
Nosocomial diarrhea is a common problem.There are multiple ethiologies of nosocomial diarrhea in which can be divided into inflammatory and non inflammatory diarrhea. Fecal calprotectin is a good marker to identify inflammatory diarrhea in outpatient setting; for example, differentiating inflammatory bowel disease and irritable bowel syndrome. Its performance in inpatient setting has not been well established. This study aim to determine the efficacy of fecal calprotectin in distinguishing inflammatory nosocomial diarrhea from non-inflammatory nosocomial diarrhea.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional, and observational study. The patients with nosocomial diarrhea whose stool samples are sent for stool examination and Clostridium difficile toxin by their treating physicians will be recruited. Their leftover stool samples will be kept at - 80 c and will be measured for calprotectin level at the end of study. The patients will be treated by their treating physicians. They will be classified into 2 groups - inflammatory and non-inflammatory diarrhea.

The inflammatory diarrhea will be defined if 1) positive for C. difficile toxin or 2) stool WBC more than 5/HPF or 3) inflammatory mucosa or ulceration noted on colonoscopy.

The noninflammatory diarrhea will be defined if 1)negative for C. difficile toxin and 2) no WBC on stool examination and 3) dramatic response to diet adjustment or 4) no mucosal inflammation or ulceration if colonoscopy is performed

The patients who do not respond to diet modification, but do not undergo colonoscopy will be excluded because the definite diagnosis cannot be made.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 hear
* Diarrhea more than 3 time per day after admitted in hospital more than 72 hours

Exclusion Criteria:

* intraabdominal pressure more than 12 mmHg
* patient on chemotherapy with neutropenia ,ANC less than 1,000/mm3
* patients whose definite diagnosis cannot be obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients in Siriraj hospital, Bangkok, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Fecal calprotectin levels | 1 day
  Compare fecal calprotectin levels in patients with inflammatory nosocomial diarrhea and non-inflammatory nosocomial diarrhea

SECONDARY OUTCOMES:
Prognosis of hospitalized patients with nosocomial diarrhea. | 30 days
  Correlation of fecal calprotectin levels and prognosis of hospitalized patients with nosocomial diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Julajak Limsrivilai, MD, MSc, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pawlowski SW, Warren CA, Guerrant R. Diagnosis and treatment of acute or persistent diarrhea. Gastroenterology. 2009 May;136(6):1874-86. doi: 10.1053/j.gastro.2009.02.072. Epub 2009 May 7. PMID 19457416
- [Background] Reintam Blaser A, Deane AM, Fruhwald S. Diarrhoea in the critically ill. Curr Opin Crit Care. 2015 Apr;21(2):142-53. doi: 10.1097/MCC.0000000000000188. PMID 25692805
- [Background] Chang SJ, Huang HH. Diarrhea in enterally fed patients: blame the diet? Curr Opin Clin Nutr Metab Care. 2013 Sep;16(5):588-94. doi: 10.1097/MCO.0b013e328363bcaf. PMID 23799327
- [Background] Bartlett JG. Clinical practice. Antibiotic-associated diarrhea. N Engl J Med. 2002 Jan 31;346(5):334-9. doi: 10.1056/NEJMcp011603. No abstract available. PMID 11821511
- [Background] Siciliano RF, Castelli JB, Randi BA, Vieira RD, Strabelli TM. Cytomegalovirus colitis in immunocompetent critically ill patients. Int J Infect Dis. 2014 Mar;20:71-3. doi: 10.1016/j.ijid.2013.11.008. Epub 2014 Jan 6. PMID 24406737
- [Background] Manabe YC, Vinetz JM, Moore RD, Merz C, Charache P, Bartlett JG. Clostridium difficile colitis: an efficient clinical approach to diagnosis. Ann Intern Med. 1995 Dec 1;123(11):835-40. doi: 10.7326/0003-4819-123-11-199512010-00004. PMID 7486465
- [Background] Crobach MJ, Dekkers OM, Wilcox MH, Kuijper EJ. European Society of Clinical Microbiology and Infectious Diseases (ESCMID): data review and recommendations for diagnosing Clostridium difficile-infection (CDI). Clin Microbiol Infect. 2009 Dec;15(12):1053-66. doi: 10.1111/j.1469-0691.2009.03098.x. PMID 19929972
- [Background] van Rheenen PF, Van de Vijver E, Fidler V. Faecal calprotectin for screening of patients with suspected inflammatory bowel disease: diagnostic meta-analysis. BMJ. 2010 Jul 15;341:c3369. doi: 10.1136/bmj.c3369. PMID 20634346
- [Background] Menees SB, Powell C, Kurlander J, Goel A, Chey WD. A meta-analysis of the utility of C-reactive protein, erythrocyte sedimentation rate, fecal calprotectin, and fecal lactoferrin to exclude inflammatory bowel disease in adults with IBS. Am J Gastroenterol. 2015 Mar;110(3):444-54. doi: 10.1038/ajg.2015.6. Epub 2015 Mar 3. PMID 25732419
- [Background] Mosli MH, Zou G, Garg SK, Feagan SG, MacDonald JK, Chande N, Sandborn WJ, Feagan BG. C-Reactive Protein, Fecal Calprotectin, and Stool Lactoferrin for Detection of Endoscopic Activity in Symptomatic Inflammatory Bowel Disease Patients: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2015 Jun;110(6):802-19; quiz 820. doi: 10.1038/ajg.2015.120. Epub 2015 May 12. PMID 25964225
- [Background] Whitehead SJ, Shipman KE, Cooper M, Ford C, Gama R. Is there any value in measuring faecal calprotectin in Clostridium difficile positive faecal samples? J Med Microbiol. 2014 Apr;63(Pt 4):590-593. doi: 10.1099/jmm.0.067389-0. Epub 2014 Jan 25. PMID 24464697
- [Background] Popiel KY, Gheorghe R, Eastmond J, Miller MA. Usefulness of Adjunctive Fecal Calprotectin and Serum Procalcitonin in Individuals Positive for Clostridium difficile Toxin Gene by PCR Assay. J Clin Microbiol. 2015 Nov;53(11):3667-9. doi: 10.1128/JCM.02230-15. Epub 2015 Sep 9. PMID 26354814
- [Background] Barbut F, Gouot C, Lapidus N, Suzon L, Syed-Zaidi R, Lalande V, Eckert C. Faecal lactoferrin and calprotectin in patients with Clostridium difficile infection: a case-control study. Eur J Clin Microbiol Infect Dis. 2017 Dec;36(12):2423-2430. doi: 10.1007/s10096-017-3080-y. Epub 2017 Aug 12. PMID 28801865
- [Background] Swale A, Miyajima F, Roberts P, Hall A, Little M, Beadsworth MB, Beeching NJ, Kolamunnage-Dona R, Parry CM, Pirmohamed M. Calprotectin and lactoferrin faecal levels in patients with Clostridium difficile infection (CDI): a prospective cohort study. PLoS One. 2014 Aug 29;9(8):e106118. doi: 10.1371/journal.pone.0106118. eCollection 2014. PMID 25170963
- [Background] Kim J, Kim H, Oh HJ, Kim HS, Hwang YJ, Yong D, Jeong SH, Lee K. Fecal Calprotectin Level Reflects the Severity of Clostridium difficile Infection. Ann Lab Med. 2017 Jan;37(1):53-57. doi: 10.3343/alm.2017.37.1.53. PMID 27834066
- [Background] Peretz A, Tkhawkho L, Pastukh N, Brodsky D, Halevi CN, Nitzan O. Correlation between fecal calprotectin levels, disease severity and the hypervirulent ribotype 027 strain in patients with Clostridium difficile infection. BMC Infect Dis. 2016 Jun 22;16:309. doi: 10.1186/s12879-016-1618-8. PMID 27334992

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT04491799/Prot_SAP_000.pdf